CLINICAL TRIAL: NCT02122783
Title: Comparison of the Functional Walking Outcomes of Two Settings of a Commercially Available Ankle Foot Orthosis in Adult Stroke Patients
Brief Title: Comparison of the Functional Walking Outcomes of Two Settings of a Commercially Available AFO in Adult Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Mukul Talaty, Biomechanist, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HN 4422
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Walking Aided by a Leg Brace in Stroke Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional then Experimental brace resistance (Experimental): Participants received the Default intervention for a period of a month, were evaluated in the lab and then the novel intervention was administered for use for the next month. There was a small period (few hours in the lab) where the subject was transitioned to the second intervention.
  Interventions: Device: ADR™ brace resistance; Device: Conventional brace resistance (using hard stops)
- Experimental then Conventional brace resistance (Experimental): Participants received the the novel elastomer to provide brace support intervention for a period of a month, were evaluated in the lab and then the conventional intervention was administered for use for the next month. There was a small period (few hours in the lab) where the subject was transitioned to the second intervention.
  Interventions: Device: ADR™ brace resistance; Device: Conventional brace resistance (using hard stops)

INTERVENTIONS:
Device: ADR™ brace resistance
Device: Conventional brace resistance (using hard stops) — Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs

SUMMARY:
The purpose of this study is to evaluate how two different settings of a commercially available ankle foot brace affect how stroke patients walk. The study brace is an ankle foot orthosis (AFO) that makes use of a newer type of joint that contains a soft insert, in addition to the conventional hard stops, to limit the range of motion of the ankle during walking. The results of this study will help to clarify 1) whether and how this new joint affects the way you walk, 2) whether it makes it easier for the clinician to align your brace and 3) your opinions about the new joint.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how two different settings of a commercially available ankle foot brace affect how stroke patients walk. The study brace is an ankle foot orthosis (AFO) that makes use of a newer type of joint that contains a soft insert, in addition to the conventional hard stops, to limit the range of motion of the ankle during walking. Participants undergo testing in the gaitlab after using the new brace for a period of time. The results of this study will help to clarify 1) whether and how this new joint affects the way you walk, 2) whether it makes it easier for the clinician to align your brace and 3) your opinions about the new joint.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 21 and 70 males and non-pregnant females
2. Diagnosis of stroke more than 1 year ago
3. Ambulatory at 0.5m/s or greater
4. Require unilateral AFOs to ambulate
5. Stable medical condition - no concomitant progressive diseases that could affect motor function
6. Ability to comply with directions and cooperate with research team

Exclusion Criteria:

1. Subjects who are currently receiving physical therapy for gait problems
2. Anticipated surgical or pharmacologic intervention for tone/contractures during the study period
3. Additional neurologic or musculoskeletal diagnoses that might impair gait (i.e., recent orthopedic interventions (6 weeks), unhealed fractures, significant degenerative joint disease, lower limb amputation, uncontrolled seizures)
4. Recent cardiac or active pulmonary disease, liable blood pressure
5. Recent back surgery

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mukul Talaty, PhD, Principal Investigator — Albert Einstein (MossRehab)
Locations (1):
- MossRehab, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross over study - so all participants received both interventions (i.e. were in both study arms).
Groups:
- Conventional Then Experimental Brace Resistance: Default intervention Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs
  Experimental intervention Same MAFO but with ADR (soft polymer) providing brace resistance
- Experimental Then Conventional Brace Resistance: Experimental Condition Using the novel elastomer (ADR™ ) to provide brace resistance
  Conventional Condition Same MAFO as above but using pins/springs to provide brace resistance
Period: Overall Study
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Conventional Then Experimental Brace Resistance: Conventional intervention Conventional brace resistance (using hard stops): Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs
  Experimental intervention Same MAFO as above but now using ADR™ soft polymer as brace resistance
- Experimental Then Conventional Brace Resistance: Experimental intervention Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing ADR™ soft polymer as brace resistance
  Conventional intervention Same MAFO as above but now using springs/pins as brace resistance
- Total: Total of all reporting groups
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (17.0) | 55.5 (3.5) | 54.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Self-selected Walking Velocity
Description: walking velocity will be assessed by an electronic temporospatial foot-fall measurement system (gaitmat)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Conventional Brace Resistance (Hardstop): Default intervention
  Conventional brace resistance (using hard stops): Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs
- ADR™ Brace Resistance: Condition using the novel elastomer to provide brace support
  ADR™ brace resistance
Arm/Group | Conventional Brace Resistance (Hardstop) | ADR™ Brace Resistance
Number analyzed (Participants) | 5 | 5
m/s | 0.71 (.39) | 0.74 (.38)

2. Primary Outcome: Step Length Symmetry
Description: step length symmetry will be assessed by an electronic temporospatial foot-fall measurement system (gaitmat). symmetry will result in a ratio of step length on more involved or affected side compared to the less involved or affected (i.e. the "normal") side. as such, the measure will appear to have no units but actually will be a ratio of the same units (in this case, meters to meters).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio (m/m)
Groups:
- Conventional Then Experimental Brace Resistance: Conventional intervention Conventional brace resistance (using hard stops): Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs
  Experimental is same MAFO but just using soft polymer inserts to provide the brace resistance
- Experimental Then Conventional Brace Resistance: Condition using the novel elastomer to provide brace support: ADR™ brace resistance
  Conventional refers to same brace but using pins/springs to provide brace resistance
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance
Number analyzed (Participants) | 2 | 3
ratio (m/m) | 0.98 (.24) | 0.96 (.25)

3. Primary Outcome: Step Time Symmetry
Description: step time symmetry will be assessed by an electronic temporospatial foot-fall measurement system (gaitmat). symmetry will result in a ratio of step time on more involved or affected side compared to the less involved or affected (i.e. the "normal") side. as such, the measure will appear to have no units but actually will be a ratio of the same units (in this case, seconds to seconds).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio (seconds/seconds)
Groups:
- Conventional Brace Resistance (Hardstop): Conventional intervention:
  Conventional polypropylene custom molded ankle foot orthosis (MAFO) with Lawrence style double channel adjustable joints containing pins/springs
  Experimental intervention:
  Same MAFO as above but with soft polymer insert to provide the brace resistance.
Arm/Group | Conventional Brace Resistance (Hardstop) | ADR™ Brace Resistance
Number analyzed (Participants) | 2 | 3
ratio (seconds/seconds) | 1.03 (.52) | 0.99 (.43)

4. Secondary Outcome: Joint Kinematics
Description: joint kinematics will be assessed using motion capture system
Time Frame: 8 weeks
Population: These data will never be analyzed as they were not collected.
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Joint Kinetics
Description: joint kinematics will be assessed using motion capture and biomechanical force measurement systems
Time Frame: 8 weeks
Population: These data will never be analyzed as they were not collected.
Arm/Group | Conventional Brace Resistance (Hardstop) | ADR™ Brace Resistance
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Activity (Step Count)
Description: activity will be measured using accelerometer based step activity monitoring devices
Time Frame: 8 weeks
Population: These data will never be analyzed as they were not collected.
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Subject Opinions
Description: subject opinions will be measured using surveys and questionnaires
Time Frame: 8 weeks
Population: These data will never be analyzed as they were not collected.
Arm/Group | Conventional Then Experimental Brace Resistance | Experimental Then Conventional Brace Resistance
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Conventional Brace Resistance (Hardstop) | ADR™ Brace Resistance
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Brace Resistance (Hardstop) (N=5) | ADR™ Brace Resistance (N=5)
discomfort while driving, back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No